CLINICAL TRIAL: NCT00439101
Title: A Randomized, Double Blind, Placebo-Controlled Trial of Megestrol Acetate as an Appetite Stimulant in Malnourished Children With Cancer
Brief Title: A Randomized Clinical Trial of Megestrol Acetate as an Appetite Stimulant in Malnourished Children With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H06-03499; CW06- 0294 (Other: Hospital Review)
Record Dates: First submitted 2007-02-21; First posted 2007-02-23 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Malnourished Children With Cancer
Keywords: weight loss; malignancy; corticosteroids; supplemental feeding; adrenal insufficiency; diabetes
MeSH Terms: conditions — Weight Loss; Neoplasms; Adrenal Insufficiency; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Megstrol Acetate
- 2 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Megstrol Acetate — Megestrol acetatet 7.5 mg/kg/day orally (lemon-lime suspension) for 90 days.
  Arms: 1
Other: Placebo — Placebo (lemon-lime suspension) taken orally for 90 days.
  Arms: 2

SUMMARY:
The purpose of this research study is to determine if megestrol acetate can be used as an appetite stimulant to improve weight gain in children with cancer and poor nutrition. The study design is a randomized, double blind, placebo controlled trial. Secondarily, we would like to determine what effect any improvement in weight has on body composition by DEXA scan. This includes whether the drug results in an increase in fat, fat-free mass, or both. If our patients gain weight we would like to know if it improves their quality of life. Finally, many children with cancer lose too much weight and require feeding to occur through a tube put down their nose into their stomach (NG feeding). The tube can be painful to put down and is uncomfortable when in. Some children may also require nutrition to be given into a vein (Total Parenteral Nutrition or TPN). We are trying to see if we can prevent these procedures from happening by having the subjects gain weight. This study will tell doctors if the drug truly works (or does not work) in children who are underweight.

DETAILED DESCRIPTION:
Overview of the study phases Prior to the randomization phase, we will draw some blood work (1 teaspoon) with regular blood work to see if you/your child meet the final eligibility requirements. If the results are within normal limits, we will proceed on to the Randomization Phase. If the results are not within normal limits for your/your child's age, then you/your child will not be able to proceed with the study and we will pass these test results on to your regular oncologist.

Randomization Phase If you/your child agree to take part in this study you/your child will have an equal chance of receiving one of two possible liquids: Megace (7.5 mg/kg/day taken once in the morning) or the same amount of a placebo (a placebo is a substance that looks and tastes exactly like the real medicine, however it is an inactive substance that contains no drug). This assigning to the drug or the placebo is called randomization. Neither you nor your physician can choose or know which treatment you are receiving. This "blinding" is necessary to fairly test these drugs. In an emergency, your physician can immediately find out which of the drugs/treatments you are receiving.

Once randomized, you/your child will be given a supply of the drug or the placebo. Both the drug and the placebo are a lemon-lime flavored liquid. There are no pills or tablets to take. You/your child are to take the liquid by mouth in the amount prescribed once per day. You will take the liquid every day for 90 days (3 months). The liquid is to be taken half an-hour before breakfast.

Pre-treatment Information Collection Phase Before you/your child start taking the liquid, we will collect some initial information. This will include taking your/your child's weight and height. A dietitian will perform an assessment of you/your child's body composition using a tool called a caliper. This will briefly pinch the skin at the back of your/your child's arm. It will not hurt. The dietitian will also measure your/your child's upper arms using a tape measure.

A research nurse will ask a series of questions called a Quality of Life assessment. This will tell us about how you/your child feels before starting the study.

Afterwards, you/your child will have a scan called a DEXA (stands for Dual Energy X-Ray Absorptiometry) scan done to assess your/your child's body composition. A DEXA scan does not hurt but requires that you/your child lie still on the table while the scanner moves over you/your child. Like all scans, there is some radiation exposure. However, the total amount of radiation is very small (about half the radiation exposure of a normal chest xray). This should not cause any problem for you/your child.

We will also draw some additional blood (approximately 1 teaspoon) from your central line. You/your child will not have extra pokes for the purposes of this study.

Follow-up Phase You/your child will be followed closely by our team of doctors and dieticians during the 90 days you/your child are on the study. Follow-up will occur when you are normally scheduled to see your doctor. This can occur at either the Pediatric Oncology outpatient clinics or when you are admitted to the BC Children's Hospital (Vancouver) or Stollery Children's Hospital (Edmonton). You do not have to make special appointments for the purpose of this study.

We will watch your weight closely during the 3 months of the study. If you/your child lose an additional 15% from your/your child's baseline (starting) weight we will stop you taking the medication or placebo. You will then receive regular medical care. This may include starting tube feeding or TPN.

We will also take additional blood work at least every 2 weeks during the 3 months. This can be done through your/your child's central line at times when regular blood work is being drawn. Once a month our research nurse will contact you by phone to see how things are going and ask questions about possible side effects.

Study Conclusion Phase At the end of the study we will again collect all the information as we did in the Pre-treatment Information Collection Phase. This will include your/your child's weight, height, caliper and arm measurements as well as asking the same quality of life questions. You will then have a second DEXA scan done.

After 90 days you will be told whether you received the drug (Megace) or the inactive substance (Placebo).

The time commitment for you/your child to take part in this research should be minimal. Each DEXA scan (you/your child are asked to complete 2 DEXA scans during the study) will take approximately 1 hour. Each study nurse interview (3) should take approximately 10-15 minutes each time. The quality of life questions will be asked three times and take approximately 5-10 minutes each time to complete.

ELIGIBILITY:
Inclusion Criteria:

1. Any subject with malnourishment presumed secondary to cancer or cancer- related therapy is eligible. Malnourishment is defined as one or more of the following at the time of enrollment on study:

   * A documented weight loss of ≥ 5% not attributable to acute fluid losses.
   * A weight deficit <90% expected for height, age and gender not attributable to acute fluid losses.
   * A mid upper-arm circumference < 5th percentile for age and gender.
2. Subjects with malignancy (except those covered in the exclusion criteria) either at diagnosis or during active therapy.
3. Subjects with relapsed disease are eligible for study.
4. Subjects on palliative therapy are eligible for study provided that the predicted life expectancy is at least 3 months.
5. Subjects must be <18 years at the time of admission to this study.
6. Subjects to receive corticosteroids while on study are eligible provided they are not required for >7 days in a 6-week period. The beginning of the 6-week period is defined as the day the first dose of corticosteroids is taken.
7. Subjects who received >7 days of corticosteroids in the previous 6-weeks before entering the study are eligible provided they have not received corticosteroids in the preceding 14 days.
8. Signed informed consent must be obtained according to institutional guidelines before enrollment on study.

Exclusion Criteria:

1. Any child receiving nutritional intervention including supplemental enteral (nasogastric / nasojejunal / gastrostomy) or parenteral (TPN) nutrition.
2. Subjects expected to receive corticosteroids for >7 days in a 6-week period. The 6-week period will be defined as starting the first day the steroids are to be taken.
3. Subjects in the previous 6-weeks who received >7 days of corticosteroids AND who are not at least 14 days from their last dose of corticosteroids.
4. Subjects concurrently prescribed other appetite-stimulating medications.
5. Subjects with hormone-sensitive tumors including meningiomas.
6. Subjects with any of the following conditions:

   * Adrenal insufficiency Defined as: A pre-study 8:00 AM serum cortisol lower than the defined limits of this study (see section 7.4) plus confirmation of adrenal insufficiency by an ACTH stimulation test.
   * Diabetes Mellitus Defined as: A pre-study random chemstrip or venous blood glucose >10 mmol/L with confirmation by a fasting blood glucose the next morning greater than the normal limits defined for this study
   * Pregnancy
   * Subjects with acute illnesses deemed clinically significant by the study coordinator (e.g., sepsis, congestive heart failure, hypertensive crises, in intensive care unit, acute or chronic renal failure, acute or chronic hepatic failure).
   * Subjects with previous or current thromboembolic conditions (excluding central venous thrombosis related to the placement of a central venous catheter).
7. Subjects with a predicted life expectancy less than 3 months.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2007-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
To determine if daily administration of megestrol acetate (MA) for 3 months compared to placebo prevents weight loss or improves weight gain in children with cancer-associated anorexia-cachexia.

SECONDARY OUTCOMES:
• To investigate whether MA results in improvement in other anthropometric measures of nutritional status (e.g. weight-for-height, triceps skinfolds, mid upper-arm circumference).
To investigate whether MA has a beneficial effect on body composition using dual-energy x-ray absorptiometry (DXA).
To determine if appetite stimulation following MA therapy results in improved quality of life for children with cancer-associated cachexia.
To determine if MA results in fewer requirements for invasive nutritional support such as tube feeding, gastrostomy tubes, and TPN.
To evaluate toxicities associated with MA in pediatric oncology subjects.

CONTACTS AND LOCATIONS:
Overall Officials: David Dix, MD, Principal Investigator — University of British Columbia; Beverly Wilson, MD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - Stollery Children's Hospital, Edmonton, British Columbia
  - Children's & Women's Health Centre of British Columbia, Vancouver, British Columbia